CLINICAL TRIAL: NCT06259968
Title: Neuromuscular Electrical Stimulation Superimposed or Not on Voluntary Contraction After Reconstruction of the Anterior Cruciate Ligament: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Bruno Manfredini Baroni, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 76203223.0.0000.5345
Record Dates: First submitted 2024-01-23; First posted 2024-02-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation; Anterior Cruciate Ligament Reconstruction
Keywords: Neuromuscular Electrical Stimulation; Knee; Physiotherapy; Quadriceps; Anterior cruciate ligament reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES+ (Experimental): Neuromuscular electrical stimulation with superimposed voluntary contraction
  Interventions: Device: Neuromuscular electrical stimulation with superimposed voluntary contraction
- NMES (Active Comparator): Neuromuscular electrical stimulation without voluntary contraction
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Patients in the neuromuscular electrical stimulation group will receive neuromuscular electrical stimulation without the concomitant execution of voluntary quadriceps contraction
  Other Names: NMES
  Arms: NMES
Device: Neuromuscular electrical stimulation with superimposed voluntary contraction — Patients will be instructed to perform maximum voluntary contractions superimposed on neuromuscular electrical stimulation
  Other Names: NMES +
  Arms: NMES+

SUMMARY:
This study aims to evaluate the effectiveness of neuromuscular electrical stimulation with superimposed voluntary contraction (NMES+ group) compared to NMES without voluntary contraction (NMES group) during the initial month of rehabilitation post anterior cruciate ligament reconstruction (ACLR). Forty patients will be randomly assigned to either the NMES group or the NMES+ group. Both groups will follow an identical rehabilitation regimen in the first month after surgery, which includes interventions for symptom management, inflammation control, edema reduction, improved joint motion range, and restoration of muscle function.

All participants will undergo identical assessment protocols at four time points: pre-surgery evaluation, and assessments at 2, 15, and 30 days post-ACLR. The primary outcome of the study is the maximal isometric strength of knee extensors. Secondary outcomes encompass thigh muscle atrophy, self-reported functional impairments, knee pain, knee edema, joint range of motion, and quadriceps activation status.

ELIGIBILITY:
Inclusion Criteria:

- Individuals of both genders, aged between 18 and 40 years, scheduled for ACL reconstruction surgery during the data collection period.

Exclusion Criteria:

* Failure to attend the pre-surgery assessment session;
* Delay of more than 7 days after surgery to initiate the rehabilitation program proposed by the study;
* Presence of injuries related to the rupture of the ACL that hinder partial weight-bearing in the first week after surgery, either due to medical recommendation or the patient inability/disposition.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal isometric strength of knee extensors | Before surgery and 30 days post-surgery.
  Assessed by manual isometric dynamometry

SECONDARY OUTCOMES:
Joint range of motion | Before surgery, and then at 2, 15, and 30 days post-surgery.
  Joint range of motion will be assessed using heel-height measurement and goniometry
Self-reported functional impairments | Before surgery, and then at 2, 15, and 30 days post-surgery.
  Self-reported functional impairments will be assessed using Lysholm Scale and the Knee Outcome Survey-Activities of Daily Living Scale (KOS-ADLS)
Quadriceps activation status | Before surgery, and then at 2, 15, and 30 days post-surgery.
  The quadriceps activation status will be assessed by lag sign.
Muscle atrophy | Before surgery, and then at 2, 15, and 30 days post-surgery.
  The evaluation of muscle atrophy will be performed by measuring the circumference of the thigh.
Knee edema | Before surgery, and then at 2, 15, and 30 days post-surgery.
  Joint swelling will be assessed using the Stroke Test.
Knee pain | Before surgery, and then at 2, 15, and 30 days post-surgery.
  The severity of knee pain will be assessed through the numerical pain rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Rehabilitation Center, Veranópolis, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No